CLINICAL TRIAL: NCT02656264
Title: The Chronic Pain Incidence After Elective and Urgent Cesarean Sections
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assistant Professor, MD, Tokat Gaziosmanpasa University
Other Study IDs: 15-KAEK-028
Record Dates: First submitted 2015-12-24; First posted 2016-01-14 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the effects of whether urgent or elective cesarean section on the occurrance of chronic pain.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of whether urgent or elective cesarean section on the occurrance of chronic pain. Patients aged between 18 - 45 years whose underwent urgent or elective cesarean section will be invited to participate in the study. Preoperatively in operating theatre, patients will be asked to complete the pain catastrophizing scale (PCS) questionnaire. In postoperative 6 months after discharge, patients will be called by an investigator who is blind to the study to evaluate the presence of chronic pain. Patients will be asked to grade the pain that they suffer using a numeric rating scale for the intensity of pain.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 - 45 years of age
* underwent elective or urgent cesarean section

Exclusion Criteria:

* not willing to participate in the study
* can not reach by phone
* use of anti-psychotic or anti-depressant drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: * Female
  * 18 - 45 years of age
  * underwent elective or urgent cesarean section
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
numeric rating scale | One time when calling the patient, an avarage of three months

SECONDARY OUTCOMES:
pain catastrophizing scale | one time in operating theatre, an avarage of three months
presence of chronic pain using numeric rating scale | One time when calling the patient, an avarage of three months

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Assist.Prof., Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided